CLINICAL TRIAL: NCT06205810
Title: Comprehensive Anatomical and Physiological Evaluation of Patients With Stable Coronary Artery Disease.
Brief Title: The COMPLETE Study
Acronym: COMPLETE
Status: Recruiting | Type: Observational
Sponsor: CoreAalst BV (Industry)
Collaborators: HeartFlow, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CA-063
Record Dates: First submitted 2023-11-28; First posted 2024-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
Keywords: FFRCT
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The COMPLETE study is a single-centre, investigator-initiated study of patients with an indication for invasive coronary angiography with CCTA performed during the diagnostic evaluation. After identifying the presence of a coronary stenosis, defined as an epicardial lesion >50% stenosis on CCTA, patients eligible for the study will be invited to participate.

The main aim of this trial is to assess the accuracy of coronary CT angiography to quantify total atheroma volume with intravascular ultrasound as reference.

Patients will be divided into 2 sub-groups:

Cohort 1: Patients with stable coronary artery disease or stabilized acute coronary syndromes with a clinical indication for invasive coronary angiography.

Cohort 2: Patients previously revascularized with a metallic stent with a clinical indication for invasive coronary angiography.

In both cohorts, patients should have undergone coronary CT angiography as part of the standard of care.

Patients included in the study will be managed according to the standard of care for the assessment of coronary artery disease. Clinical follow-up will be collected until 3 years follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Epicardial stenosis more than 50% by visual assessment.

Exclusion Criteria:

1. STEMI.
2. Hemodynamic instability.
3. Rapid atrial fibrillation, flutter or arrhythmia (HR > 80 bpm).
4. Insufficient CCTA image quality.
5. Age <18 years.
6. Chronic obstructive pulmonary disease.
7. Contraindication to adenosine.
8. NYHA class III or IV, or last known left ventricular ejection fraction <30%.
9. Uncontrolled or recurrent ventricular tachycardia.
10. History of recent stroke (≤90 days).
11. Prior myocardial infarction.
12. History of ischemic stroke (>90 days) with modified RANKIN score ≥ 2.
13. History of any hemorrhagic stroke.
14. Previous coronary artery bypass surgery.
15. Active liver disease or hepatic dysfunction, defined as AST or ALT > 3 times the ULN.
16. Severe renal dysfunction, defined as an eGFR <30 mL/min/1.73 m2.
17. BMI >35 kg/m2.
18. Nitrate intolerance
19. Contra-indication to heart rate lowering drugs.
20. Unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Coronary Artery Disease with an epicardial stenosis of more than 50% of visual assessment.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2030-10-15 (Estimated); Study Completion 2031-10-15 (Estimated)

PRIMARY OUTCOMES:
assess the accuracy of CCTA to quantify total atheroma volume (TAV) with IVUS as reference. | day 0 (day of the procedure)
  To assess the accuracy of CCTA (Coronary Computed Tomography Angiography) to quantify total atheroma volume (TAV) with IVUS (Intravascular Ultrasound) as reference.

SECONDARY OUTCOMES:
Assess the accuracy of CCTA to determine minimal stent area with IVUS as reference. | day 0 (day of the procedure)
  To assess the accuracy of CCTA (Coronary Computed Tomography Angiography) to determine minimal stent area with IVUS (Intravascular Ultrasound) as reference.
Determine the diagnostic performance (mean difference) of FFRCT in stented segments with invasive FFR as reference. | day 0 (day of the procedure)
  To determine the diagnostic performance (mean difference) of FFRCT (Fractional Flow Reserve derived from CT) in stented segments with invasive FFR (Fractional Flow Reserve ) as reference.
Describe the impact of coronary microvascular dysfunction assessed by IMR and absolute coronary resistance on the accuracy of FFRCT. | day 0 (day of the procedure
  To describe the impact of coronary microvascular dysfunction assessed by IMR (Index of Microcirculatory Resistance) and absolute coronary resistance on the accuracy of FFRCT (Fractional Flow Reserve derived from CT).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wyffels, MD, PhD, Principal Investigator — OLV Hospital Aalst
Locations (1):
- OLV Hospital Aalst, Aalst, Oost-Vlaanderen, Belgium